CLINICAL TRIAL: NCT03699787
Title: The Effects of a Graphomotor Intervention Program According to a Psychomotor Approach on Graphomotor Competences in Preschool Children: A Randomized Controlled Trial
Brief Title: Graphomotor Intervention Program for Handwriting Difficulties Prevention in Preschool Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Helena Isabel Falcão Coradinho, Principal Investigator, University of Évora
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 05102018
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Typical Development; Risk of Dysgraphia; Dysgraphia
Keywords: Graphomotor intervention program; Preschool children; Graphomotor competences; Prevention
MeSH Terms: conditions — Agraphia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graphomotor intervention program (Experimental): The experimental group (EG) intervention comprises a graphomotor intervention program according to a psychomotor approach. The program integrates two group sessions (6-8 children)/week of 30 minutes for 8 weeks (16 sessions).
  Interventions: Other: Graphomotor intervention program
- Control Group (No Intervention): The control group (CG) participants will maintain their normal classroom activities. After the study, control group participants will be offered the opportunity to integrate a similar graphomotor intervention program.

INTERVENTIONS:
Other: Graphomotor intervention program — The graphomotor intervention program aims to promote the development and reinforcement, different skills involved in the learning process of handwriting and has a preventive character. It follows a bodily, playful, multisensory, exploratory (sensory integration) and neuromotor task training approach and focuses on the following intervention domains: segmental awareness, passive relaxation, trunk-limb dissociation, interdigital coordination, attention, planning, spatial organization/orientation and perception.
  Arms: Graphomotor intervention program

SUMMARY:
12-30% of children present handwriting difficulties, which has negative repercussions on their school career. For this reason, it is fundamental to bet on their prevention. The aim of present study is to examine the effects of a graphomotor intervention program on graphomotor competences in children in the last year of preschool education. This experimental study is a randomized controlled trial. The program will run for 8 weeks (2 sessions/week of 30 minutes), followed by 6 months of follow-up without intervention. Participants will be assessed 1) at baseline, 2) at the end of the program, and 3) after the follow-up. Participants will be randomly allocated to two groups: experimental group (graphomotor intervention program) and control group.

DETAILED DESCRIPTION:
According to estimates, 12 to 30% of children have handwriting difficulties (1), which has negative consequences for school success (2). In addition, this is one of the main reasons for referral and consultation in psychomotricity in school-age (3), which reflects the urgency of acting in this field.

The need for prevention and early intervention is indisputable (4). Several studies indicate that both outweigh the benefits of late intervention, because as time goes on it is increasingly difficult to correct handwriting difficulties (5-6).

Graphomotor skills include the trait, the drawing and the formal handwriting and are related to long and complex learning, which requires several years of learning (7-9).

Today it is known that preschool education represents a very important period for the development of these skills (10). In preschool, children spend 42% of the day on paper and pencil tasks (11) and it is during this period that handwriting readiness skills are developed (12), being a predictor of future school success (12-15). For Beery (16) children are not apt to learn to handwrite without first copying the first nine figures of the Beery-Buktenica Developmental Test of Visual-Motor Integration (VMI).

It is based on this that intervention programs have been developed with the aim of promoting the development of handwriting readiness skills in preschool age and of preventing possible handwriting difficulties at school age (14, 17). These intervention programs have shown favourable results in improving the graphomotor skills of preschool children (12, 17-18).

In most cases only something is done, once the handwriting difficulties are installed. In addition, there are few studies dedicated to intervention in graphomotor skills at preschool age and to my knowledge, there is no study whose intervention is based on a psychomotor approach. Based on this, a graphomotor intervention program with a psychomotor approach was developed, by Matias and Vieira (19), who will apply in this study to children in the last year of preschool education.

ELIGIBILITY:
Inclusion Criteria:

* Children in the last year of preschool education (aged 5 years old);
* Participation agreement.

Exclusion Criteria:

* Diagnosed or suspected of neurological disabilities (e.g., cerebral palsy, epilepsy), psychiatric and/or behavioural disorders;
* Presence of uncorrected vision and hearing problems;
* Referenced by Special Education/National Service of Early Intervention in Childhood;
* Native language is not Portuguese;
* Children with direct intervention in graphomotor skills or who had a similar intervention to that proposed less than 1 year ago;
* Participation in the intervention program of less than 80%;
* Children undergoing drug therapy (e.g., antihistamines) that interfere with the study variables;
* Do not wish to participate in the study.

Ages: 5 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline, between and within groups comparison, in Manual Preference | 0, 4, 10 months
  Outcome Measure - Manual Preference Questionnaire to assess manual preference
Change from Baseline, between and within groups comparison, in Motor Performance | 0, 4, 10 months
  Outcome Measure - Movement Assessment Battery for Children - Second Edition to assess manual dexterity, aiming and catching and balance
Change from Baseline, between and within groups comparison, in Visual-Motor Integration | 0, 4, 10 months
  Outcome Measure - Beery-Buktenica Developmental Test of Visual-Motor Integration, Sixth Edition to assess visual-motor integration, visual perception and motor coordination
Change from Baseline, between and within groups comparison, in Computerized Handwriting Process Measures | 0, 4, 10 months
  Outcome Measure - The MovAlyzeR to assess spatial, temporal and kinematic variables of handwriting

SECONDARY OUTCOMES:
Sociodemographic characteristics | 0 months
  The Sociodemographic Questionnaire collects data on the identification of the child, the parents, the sociodemographic context and the socioeconomic status of the family based on the Graffar Social Classification Scale Adapted

CONTACTS AND LOCATIONS:
Overall Officials: Helena IF Coradinho, MSc, Principal Investigator
Locations (1):
- Helena Isabel Falcão Coradinho, Evora, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alhusaini AA, Melam GR, Buragadda S. Short-term sensorimotor-based intervention for handwriting performance in elementary school children. Pediatr Int. 2016 Nov;58(11):1118-1123. doi: 10.1111/ped.13004. Epub 2016 Jul 7. PMID 27085075
- [Background] Soppelsa R, Albaret JM. Caractéristiques de la dysgraphie ou du trouble de l'apprentissage de la graphomotricité (TAG) au collège. A.N.A.E. 2014 Fev; 128:1-6. Available at: http://www.psychomot.ups-tlse.fr/Soppelsa-Albaret2014.pdf
- [Background] Lachaux-Parker C. Troubles de l'écriture et psychomotricité. Revue francophone d'orthoptie. 2012; 5:143-7. doi: 10.1016/j.rfo.2013.02.002
- [Background] Borghese NA, Palmiotto C, Essenziale J, Mainetti R, Granocchio E, Molteni B et al. Assessment of Exergames as Treatment and Prevention of Dysgraphia. In: Ibáñez J, González-Vargas J, Azorín J, Akay M, Pons J. Converging Clinical and Engineering Research on Neurorehabilitation II. Cham: Springer; 2017. p. 431-6.
- [Background] Graham S, Harris KR. Preventing Writing Difficulties: Providing Additional Handwriting and Spelling Instruction to At-Risk Children in First Grade. Teaching Exceptional Children. 2006 May/Jun; 38(5):64-66. doi: 10.1177/004005990603800509
- [Background] Graham S, Harris KR, & Fink B. Is handwriting causally related to learning to write? Treatment of handwriting problems in beginning writers. Journal of Educational Psychology. 2000; 92(4):620-33. doi: 10.1037/0022-0663.92.4.620
- [Background] Feder KP, Majnemer A. Handwriting development, competency, and intervention. Dev Med Child Neurol. 2007 Apr;49(4):312-7. doi: 10.1111/j.1469-8749.2007.00312.x. PMID 17376144
- [Background] Morin MF, Bara F, Alamargot D. Apprentissage de la graphomotricité à l'école: Quelles acquisitions? Quelles pratiques? Quels outils?. Scientia Paedagogica Experimentalis. 2017 Jul; 54(1-2):47-84. Available at: https://researchgate.net/publication/204380193_Apprentissage_de_la_graphomotricite_a_l'école_Quelles_acquisitions_Quelles_pratiques_Quels_outils
- [Background] Zeziger P, Deonna T, Mayor C. L'acquisition de l'écriture. Enfance. 2000; 3:295-304. Available at: http://www.persee.fr/doc/enfan_0013-7545_2000_num_53_3_3186
- [Background] Puranik CS, Lonigan CJ. From Scribbles to Scrabble: Preschool Children's Developing Knowledge of Written Language. Read Writ. 2011 May;24(5):567-589. doi: 10.1007/s11145-009-9220-8. PMID 22448101
- [Background] Marr D, Cermak S, Cohn ES, Henderson A. Fine motor activities in Head Start and kindergarten classrooms. Am J Occup Ther. 2003 Sep-Oct;57(5):550-7. doi: 10.5014/ajot.57.5.550. PMID 14527117
- [Background] Lifshitz N, Har-Zvi S. A Comparison Between Students Who Receive and Who Do Not Receive a Writing Readiness Interventions on Handwriting Quality, Speed and Positive Reactions. Early Childhood Educ J. 2014 Jan; 43(1):47-55. doi: 10.1007/s10643-013-0629-y
- [Background] Dinehart L. Handwriting in early childhood education: Current research and future implications. Journal of Early Childhood Literacy. 2015 Mar; 15(1):97-118. doi: 10.1177/1468798414522825
- [Background] Donica D, Goins A, Wagner L. Effectiveness of Handwriting Readiness Programs on Postural Control, Hand Control, and Letter and Number Formation in Head Start Classrooms. Journal of Occupational Therapy, Schools, & Early Intervention. 2013 Dec; 6(2):81-93. doi: 10.1080/19411243.2013.810938
- [Background] van Hartingsveldt MJ, De Groot IJ, Aarts PB, Nijhuis-Van Der Sanden MW. Standardized tests of handwriting readiness: a systematic review of the literature. Dev Med Child Neurol. 2011 Jun;53(6):506-15. doi: 10.1111/j.1469-8749.2010.03895.x. Epub 2011 Feb 11. PMID 21309763
- [Background] Beery KE. The Developmental Test of Visual/Motor Integration. CJeveland: Modern Curriculum Press; 1982.
- [Background] Spanaki I, Venetsanou F, Evaggelinou C, Skordilis E. Graphomotor skills of Greek kindergarten and elementar school children: effect of a fine motor intervention program. Comprehensive Psychology. 2014 Jan; 2(3):1-10. doi: 10.2466/01.09.IT.3.2
- [Background] Lust CA, Donica DK. Effectiveness of a handwriting readiness program in head start: a two-group controlled trial. Am J Occup Ther. 2011 Sep-Oct;65(5):560-8. doi: 10.5014/ajot.2011.000612. PMID 22026324
- [Background] Matias A, Vieira C. Programa de intervenção grafomotora. [In press].